CLINICAL TRIAL: NCT06434337
Title: Evaluation of a Novel Point-of-Care Diagnostic Test for Human Papillomavirus (HPV)
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0020; NCI-2024-04598 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Human Papillomavirus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Research Group: Standard-of-care (SOC) procedures will be performed as part of the routine visit, and the provider will collect up to two additional cervical swabs for research. One research cervicovaginal swab may also be self-collected by the patient (optional procedure) in the clinic during the routine visit. All research swab samples, in addition to residual material from standard of care HPV testing, will be transferred to Rice University team for testing and some will be tested on site at the provider facility as described below.
  Interventions: Diagnostic Test: Novel point-of-care diagnostic test for detecting HPV ("Rice HPV test")

INTERVENTIONS:
Diagnostic Test: Novel point-of-care diagnostic test for detecting HPV ("Rice HPV test") — Given by Diagnostic Test

SUMMARY:
To learn if new HPV tests can provide the same results as standard HPV tests. The findings from this study may aid in the development of new HPV tests that require less equipment and are more accessible.

DETAILED DESCRIPTION:
Primary Objectives

1. To evaluate the performance of 3 versions of a novel point-of-care diagnostic test for detecting HPV ("Rice HPV test").

Secondary Objectives

1. To evaluate the results of the Rice HPV test with corresponding pathology results to assess the association of HPV test results with the presence of high-grade cervical dysplasia (CIN 2+).
2. To assess how different sample processing methods affect the performance of the Rice HPV test.
3. To assess how different test readout methods affect the performance of the Rice HPV test.

Exploratory Objectives

1. Compare the performance of the Rice HPV test between provider-collected and self-collected samples.
2. Conduct a survey on participant experiences with self-sampling to assess whether participants prefer self-sampling over provider-collected sampling.
3. Compare the performance of the Rice HPV test to other benchmark HPV tests such as GeneXpert.

ELIGIBILITY:
Inclusion Criteria:

1. People with a cervix 21 years of age or older.
2. Scheduled to undergo hrHPV testing at MD Anderson and The Harris Health System (LBJ Hospital) according to national and institutional guidelines at time of enrollment OR are anticipated to undergo a LEEP, ECC, or biopsy.
3. Willing and able to provide informed consent.
4. Able to perform protocol-required activities. Able to speak and read English or Spanish.

Exclusion Criteria

1. Patient or provider decision not to perform HPV testing. This does not apply to patients that are undergoing either a LEEP, ECC or biopsy.
2. Participant or provider decision not to collect a sample for this study.
3. Participants that are pregnant.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Novel point-of-care diagnostic test for detecting HPV ("Rice HPV test") | Through study completion; an average of 1 year
  To evaluate the performance of the 3 version of a novel point-of-care diagnostic test for detecting HPV ("Rice HPV test").

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Schmeler, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org